CLINICAL TRIAL: NCT04589767
Title: Validation Study of the "CORNELL ASSESSMENT PEDIATRIC DELIRIUM" (CAPD)" Scale in Italian Language
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, angela amigoni, MD, Azienda Ospedaliera di Padova
Other Study IDs: 4792/AO/19
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Delirium
Keywords: delirium; monitoring
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children admitted in PICU: children enrolled will be evaluated by two nurses using CAPD Italian version. One nurse will repeat the evaluation two minutes later.
  Interventions: Behavioral: CAPD scale

INTERVENTIONS:
Behavioral: CAPD scale — Two nurses will apply CAPD scale. One nurse will repeat the CAPD evaluation two minutes later

SUMMARY:
70 children (based on the inclusion and exclusion criteria described above) admitted in PICU will be daily assessed by two nurses (inter-evaluator agreement) using the Italian version of CAPD scale administered twice at a distance of 2 minutes (intra-evaluator agreement).

DETAILED DESCRIPTION:
The psychometric validation study will take place in the PICU of the Hospital of Padua. CAPD translation and cultural adaptation was developed within the Pediatric Cardiac Surgery Intensive Care Unit of the Federico II Polyclinic.

In this study we aim to perform the psychometric validation. 70 children (based on the inclusion and exclusion criteria described above) admitted in PICU will be daily assessed by two nurses (inter-evaluator agreement) using the Italian version of CAPD scale administered twice at a distance of 2 minutes (intra-evaluator agreement).

The score will be recorded in a data collection card, all the cards will be collected and then analyzed.

ELIGIBILITY:
Inclusion Criteria:

* PICU admission
* Comfort Behavioral Score > 11

Exclusion Criteria:

* use of neuromuscular blocking agents at the moment of CAPD evaluation
* Comfort Behavioral Score < 11

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted in PICU
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
inter-evaluator agreement | 1 hour during PICU stay
  CAPD evaluation by two operators
intra-evaluator agreement | 2 minutes during PICU stay
  CAPD evaluation by two operators

CONTACTS AND LOCATIONS:
Overall Officials: angela amigoni, Principal Investigator — University Hospital Padova
Locations (1):
- PICU University Hospital of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No